CLINICAL TRIAL: NCT03919851
Title: Physician Administered Antibiotics in a Prehospital Mobile Emergency Care Unit
Brief Title: Physician Administered Antibiotics in a Prehospital Setting
Acronym: PANTIPS
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Soren Mikkelsen, Professor, Odense University Hospital
Other Study IDs: Prehospital antibiotics
Record Dates: First submitted 2019-04-16; First posted 2019-04-18 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Sepsis
Keywords: Prehospital recognition and treatment
MeSH Terms: conditions — Sepsis | interventions — Anti-Bacterial Agents; Blood Culture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Antibiotics — Administration of antibiotics
  Other Names: Blood culture

SUMMARY:
Sepsis is estimated to affect more than 30 million people globally. Detecting sepsis is notoriously difficult and there are no systems in place utilize prehospitally. In Denmark, the Mobile Emergency Care Unit (the MECU), manned by a physician and paramedic, is able to draw blood cultures and take venous lactate measurements before administering antibiotics.

This study aims to conduct a quality control on the ability of the MECU to recognize and treat sepsis by confirming the amounts of in-hospitally diagnosed cases. Furthermore the study investigates whether the blood cultures falls within an acceptable range of contamination.

DETAILED DESCRIPTION:
In Denmark, the Emergency Medical System (EMS) consists of not only ambulances operated by paramedics and emergency technicians (EMTs) but also of Mobile Emergency Care Unit (MECU) staffed with an emergency physician with specialist training in anesthesiology and a paramedic. Only the physician on the MECU can administer prehospital antibiotics in Denmark; this emphasizes the importance of the first responding emergency units' capability in detecting and realizing the need for antibiotics in a patient so that the MECU can be requested and treatment initiated quickly.

Determining the administration of antibiotics is done at the anesthesiologists' discretion.

The purpose of administering antibiotics prehospitally is to reduce the time gap between suspicion of sepsis arises and the administration of antibiotics.

The purpose of this retrospective study is to conduct a quality control of the obtaining of blood cultures and of the administration of antibiotics in the prehospital setting serviced by the MECU in Odense in the Region of Southern Denmark in a time interval of 5 years (November 2013- October 2018).

The primary purpose is to associate the prehospital tentative diagnosis (assigned by the MECU) with the final diagnosis (ICD10 from hospital charts) including: 1: An indication for antibiotic therapy and 2: An assessment of the feasibility and potential benefit of the blood cultures obtained. 3: A description of the bacteria found in the blood cultures.

The association between initial prehospital diagnosis and final the diagnosis will be compared.

Secondly the patients seen by the MECU will be characterized regarding diagnosis (ICD10-classification), age, sex, medication, and the first set of vital parameters (Heart rate, Blood pressure, Respratory rate, Oxygen saturation, Glasgow Coma Score, Temperature).

Hypothesis The indication for giving prehospital antibiotics is supported by the prehospital blood culture and by additional findings reproduced inhospitally.

The prehospital tentative diagnosis is confirmed in-hospitally. Prehospital blood sampling is associated with an acceptably low range of contamination.

ELIGIBILITY:
Inclusion: Criteria: Antibiotics administrated by prehospital physician

Exclusion: Criteria: Age below 18 years. No prehospital administration of antibiotics. Patients without inhospital medical records or patients released at the prehospital scene following treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated by the MECU in Odense from November 1st 2013 to October 31st 2018
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Prehospital diagnosis confirmed | Up to 30 days
  Prehospital tentative diagnosis matches inhospital diagnosis

SECONDARY OUTCOMES:
Blood culture positive | First day of admission
  Findings in the blood culture supports the diagnosis sepsis
Blood culture contamination below 5% | 6 days
  Findings of bacteria attributed to contamination below 1 in 20 cultures

CONTACTS AND LOCATIONS:
Locations (1):
- Mobile Emergency Care Unit in Odense, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data may be shared on reasonable request

REFERENCES:
- [Result] Perner A, Lassen AT, Schierbeck J, Storgaard M, Reiter N, Benfield T. [Disease burden and definition of sepsis in adults]. Ugeskr Laeger. 2018 Apr 9;180(15):V09170685. Danish. PMID 29690984
- [Result] Seymour CW, Kahn JM, Martin-Gill C, Callaway CW, Yealy DM, Scales D, Angus DC. Delays From First Medical Contact to Antibiotic Administration for Sepsis. Crit Care Med. 2017 May;45(5):759-765. doi: 10.1097/CCM.0000000000002264. PMID 28234754
- [Result] Moore C, Bulger J, Morgan M, Driscoll T, Porter A, Islam S, Smyth M, Perkins G, Sewell B, Rainer T, Nanayakkara P, Okolie C, Allen S, Fegan G, Davies J, Foster T, Francis N, Smith FG, Ellis G, Shanahan T, Howe R, Snooks H. Prehospital recognition and antibiotics for 999 patients with sepsis: protocol for a feasibility study. Pilot Feasibility Stud. 2018 Mar 12;4:64. doi: 10.1186/s40814-018-0258-8. eCollection 2018. PMID 29564147
- [Result] Smyth MA, Brace-McDonnell SJ, Perkins GD. Impact of Prehospital Care on Outcomes in Sepsis: A Systematic Review. West J Emerg Med. 2016 Jul;17(4):427-37. doi: 10.5811/westjem.2016.5.30172. Epub 2016 Jul 5. PMID 27429693
- [Result] Guerra WF, Mayfield TR, Meyers MS, Clouatre AE, Riccio JC. Early detection and treatment of patients with severe sepsis by prehospital personnel. J Emerg Med. 2013 Jun;44(6):1116-25. doi: 10.1016/j.jemermed.2012.11.003. Epub 2013 Jan 13. PMID 23321295
- [Result] Joynes EL, Martin J, Ross M. Management of Septic Shock in the Remote Prehospital Setting. Air Med J. 2016 Jul-Aug;35(4):235-8. doi: 10.1016/j.amj.2016.04.001. Epub 2016 May 24. PMID 27393760
- [Result] Bodilsen J, Dalager-Pedersen M, Schonheyder HC, Nielsen H. Time to antibiotic therapy and outcome in bacterial meningitis: a Danish population-based cohort study. BMC Infect Dis. 2016 Aug 9;16:392. doi: 10.1186/s12879-016-1711-z. PMID 27507415
- [Result] Andersson H, Axelsson C, Larsson A, Bremer A, Gellerstedt M, Bang A, Herlitz J, Ljungstrom L. The early chain of care in bacteraemia patients: Early suspicion, treatment and survival in prehospital emergency care. Am J Emerg Med. 2018 Dec;36(12):2211-2218. doi: 10.1016/j.ajem.2018.04.004. Epub 2018 Apr 5. PMID 29653787
- [Result] Justesen US, Larsen BW, Eshoj O, Sogaard P. [Blood cultures--indication and antibiotic therapy]. Ugeskr Laeger. 2003 May 5;165(19):1989-94. Danish. PMID 12795074